CLINICAL TRIAL: NCT03353480
Title: AN OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 3-WAY CROSSOVER BIOEQUIVALENCE STUDY COMPARING AZITHROMYCIN 250 MG TABLET (MANUFACTURED AT PFIZER DALIAN, CHINA) WITH AZITHROMYCIN 250 MG TABLET (MANUFACTURED AT PFIZER BARCELONETA, UNITED STATES) UNDER FASTED AND FED CONDITIONS IN HEALTHY CHINESE SUBJECTS
Brief Title: Bioequivalence (BE) Study Comparing Azithromycin 250 mg Tablet Manufactured in China and in the United States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0661212
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Bioequivalence
Keywords: Azithromycin tablet, Bioequivalence, Phase I, Chinese, Healthy Subjects

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, single-dose, 3-way crossover, reference scaled bioequivalence study under fasted and fed conditions in healthy Chinese subjects.
  Under each condition, subjects will be randomized to one of the 3 treatment sequences. Each treatment sequence will consist of 3 periods, separated by a washout period of at least 14 days between each period. For sequence 1, first localized originator, then originator and finally originator will be administered. The order for sequence 2 is originator, localized originator and originator. The order for sequence 3 is originator, originator and localized originator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reference (Other): 250mg Azithromycin tablet manufactured at Pfizer Barceloneta, Puerto Rico, US
  Interventions: Drug: Azithromycin Tablet manufactured in US
- Experimental (Experimental): 250mg Azithromycin tablet manufactured at Pfizer Dalian, China
  Interventions: Drug: Azithromycin Tablet manufactured in China

INTERVENTIONS:
Drug: Azithromycin Tablet manufactured in China — 250 mg Azithromycin Tablet manufactured in China
  Other Names: The localized originator, Experimental
  Arms: Experimental
Drug: Azithromycin Tablet manufactured in US — 250 mg Azithromycin Tablet manufactured in US
  Other Names: The originator, Reference
  Arms: Reference

SUMMARY:
China Food and Drug Administration (CFDA) initiated a generic consistency evaluation program to evaluate the quality and efficacy of the products manufactured in China in 2016. This is a reference scaled bioequivalence study to support the program and to demonstrate the bioequivalence between the 250 mg azithromycin tablet manufactured at Pfizer Dalian, China (the localized originator, Test) and the 250 mg azithromycin tablet manufactured at Pfizer Barceloneta, Puerto Rico, US (the originator, Reference) in healthy Chinese subjects under fasted and fed conditions. This open-lable, randomized, single-dose 3-way crossover study will enroll approximately 33 subjects for each condition. The primary endpoints are azithromycin area under the serum concentration-time curve from time zero to 72 hours post-dose (AUC72) and Cmax.

DETAILED DESCRIPTION:
This is a reference scaled bioequivalence study to support a generic consistency evaluation program, initiated by CFDA in 2016, for the evaluation of quality and efficacy of the products manufactured in China. The selected strength of 250 mg tablet is the approved strength. The primary objective is to demonstrate the bioequivalence between the 250 mg azithromycin tablet manufactured at Pfizer Dalian, China (the localized originator, Test) and the 250 mg azithromycin tablet manufactured at Pfizer Barceloneta, Puerto Rico, US (the originator, Reference) in healthy Chinese subjects under fasted (Group 1) and fed (Group 2) conditions. Approximately 33 Chinese healthy subjects will be enrolled for each group.

The primary endpoints are azithromycin area under the serum concentration-time curve from time zero to 72 hours post-dose (AUC72) and Cmax.

The secondary objective is to evaluate the safety and tolerability of azithromycin administered as a single oral dose of 250 mg tablet manufactured at Pfizer Dalian, China and 250 mg tablet manufactured at Pfizer Barceloneta, Puerto Rico, US in healthy Chinese subjects under fasted and fed conditions. And the secondary endpoint is adverse events (AEs). Other endpoints include Tmax of azithromycin, safety laboratory tests and vital signs.

In each group, subjects will be randomized to one of the 3 treatment sequences. Each treatment sequence will consist of 3 periods, separated by a washout period of at least 14 days between each period.

On Day 1 of each period in both groups, each subject will be administered investigational product at approximately 8:00 AM (± 2 hours). Blood samples for the analysis of azithromycin in serum will be collected at pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 and 72 hours post dose in each period. Vital signs, physical examination, laboratory tests and 12-lead electrocardiogram (ECG) will be performed at specified times. Tolerability and safety will be assessed for all treatments by monitoring AEs.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Healthy Chinese male and female subjects, between the ages of 18 and 45 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12-lead ECG, or clinical laboratory tests.
2. BMI of 18 to 28 kg/m2; and a total body weight ≥50 kg for males and ≥45 kg for females.
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Subjects must be of Chinese ethnicity (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent).

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen, history of drug abuse within the past 5 years.
4. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 100 mL of wine or 285 mL of beer or 25 mL of hard liquor) within 3 months of Screening.
5. Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day within 3 months prior to Screening.
6. Treatment with an investigational drug within 3 months preceding the first dose of investigational product.
7. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
8. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS complex >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
9. Female subjects of childbearing potential and fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
10. Female subjects who are breastfeeding or with positive pregnancy test at Screening and during the study period.
11. Use of prescription or nonprescription drugs, dietary supplements and herbal medicines within 14 days prior to Screening. As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor. Taking any medicinal product that changes the activity of hepatic enzymes within 28 days prior to Screening, such as a strong CYP3A4 inducer (eg, St. John's Wort).
12. Blood donation (excluding plasma donations) or loss of blood of approximately 450 mL or more within 3 months prior to Screening.
13. History of hypersensitivity to azithromycin or any components of its formulation.
14. Use of special diet (including dragon fruit, mango, citrus, etc.), strenuous activities or other factors that may affect the disposition of the study medication within 14 days prior to Screening.
15. Use of chocolate, food or beverages containing caffeine or xanthine within 48 hours prior to dosing.
16. Use of products containing alcohol within 48 hours prior to dosing.
17. Intolerance of the standard high fat breakfast, which is only applicable to the subjects participating in Group 2 (fed condition).
18. History of HIV, hepatitis B, or hepatitis C; positive testing for HIV, HepBsAg, HepBcAb, HCVAb, or TPPA.
19. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section.
20. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
21. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
AUC0-72 | 0-72 hours
  Area under the serum concentration-time profile from time zero to 72 hours post dose based on observed serum concentrations at time points 0 (prior-dose), 0.5, 1, 2, 3, 4, 5, 6,8, 10, 12, 24, 48 and 72 hours after dose using linear/log trapezoidal methods
Cmax | 0-72 hours
  Maximum serum concentration among observed serum concentrations at time points 0 (prior-dose), 0.5, 1, 2, 3, 4, 5, 6,8, 10, 12, 24, 48 and 72 hours after dose

SECONDARY OUTCOMES:
Adverse Events | Day 1 to Day 32 or early termination, plus at least 28 calendar days and up to 35 calendar days after the last administration of the investigational product
  All observed or volunteered safety events regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported during study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- The First Hospital of Jilin University/Phase I Clinical Trials Unit, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661212&StudyName=An+Open-label%2C+Randomized%2C+Single-dose%2C+3-way+Crossover+Bioequivalence+Study+Comparing+Azithromycin+250+Mg+Tablet+%28manufactured+At+Pfizer+Dalian%2C+China%29+With+Azithromycin+250+Mg+Tablet+%28manufactured+At+Pfizer+Barceloneta%2C+United+States%29+Under+Fasted+And+Fed+Conditions+In+Healthy+Chinese+Subjects